CLINICAL TRIAL: NCT03877328
Title: BioTechCOACH-ForALL: Development of Mental and Physical Exercise Systems, Clinical Recording, Supervisory Analytical Large-scale Data and Virtual Guidance of Vulnerable Population Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MIS5005517
Record Dates: First submitted 2019-02-19; First posted 2019-03-15 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: heart failure; exercise; life coach
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Coach (Experimental): BiotechCoachForAll
  Interventions: Other: BiotechCoachForAll

INTERVENTIONS:
Other: BiotechCoachForAll — A group of thirty subjects diagnosed with heart failure (HF) of any etiology undergo an experimental procedure in the following order: resting-state (eyes-closed), passively viewing thirty two agents which are grouped with respect to different appearance characteristics and passively viewing combinations of virtual agents. During the experiment, brain activity, heart rate, skin conductance, temperature and eye-gaze biosignals are collected by means of electroencephalography, Empatica E4 and Gazepoint. Subsequently, a prospective cohort study is performed in a subgroup of ten participants which undergo a three additive stage procedure. Stage 1, a wearable monitoring device (Wavelet Health) is given in order to provide objective information on the patient's activity. Stage 2, the FitForAll physical exercise program is introduced. Stage 3, introduces the coaching aspects, where personalized recommendations and suggestions are delivered through home surfaces' projection.

SUMMARY:
This would be a single center, parallel, two group randomized controlled pilot study that is designed to assess the feasibility and efficacy of the Virtual Coach Program in elderly patients with heart failure.

DETAILED DESCRIPTION:
This would be a single center, parallel, two group randomized controlled pilot study that is designed to assess the feasibility and efficacy of the Virtual Coach Program in elderly patients with heart failure. Sixteen (16) subjects will be enrolled to allow 8 subjects to be randomly assigned to each arm. The study will be conducted in Thessaloniki/Greece. The study is expected to complete enrollment in approximately 3 months. Participants will be randomly randomized to either the intervention group (use of Virtual Coach program and usual care) or the control group (use of usual care alone) after successfully fulfilling all inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged >55 years old with any of the following conditions, diagnosed according to appropriate international guidelines criteria

   a) Heart failure of any etiology, with either reduced or preserved ejection fraction
2. Subjects must be in WHO Functional Class II-IV
3. Subjects must be on stable clinical condition and on stable medical treatment for the underlying disease for at least three months prior to randomization
4. Willing and able to comply with scheduled visits, treatment plan, and trial procedures
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Patients with heart conditions other that those listed above
2. Subjects who have unstable disease with evidence of decompensation, recent hospitalization or undergoing investigation for clinical deterioration
3. Subjects with recent history of chest pain, palpitations, lightheadedness, dizziness, or syncope on exertion
4. Subjects with contraindications to physical activity or with physical obstruction to perform the prescribed training program (eg patients confined on wheel chair etc)
5. Subjects with any severe acute or chronic medical or psychiatric condition that may increase the risk associated with trial participation or may interfere with the interpretation of trial results
6. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator
7. Subjects participating in any other experimental studies
8. Subjects not willing to provide signed informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The subjects' functionality assessed both prior intervention and at the end of the study | 3 months
  Functional capacity assessed by WHO functional class
The subjects' exercise intolerance assessed both prior intervention and at the end of the study | 3 months
  Exercise intolerance assessed by distance walked in six-minute walk test
The subjects' quality of life assessed both prior intervention and at the end of the study | 3 months
  Health related quality of life assessed with the use of properly weighed for the Greek language questionnaires
  -SF-36 questionnaire
The subjects' quality of life assessed both prior intervention and at the end of the study | 3 months
  Health related quality of life assessed with the use of properly weighed for the Greek language questionnaires
  -Dukes questionnaire
Hospitalization | 3 months
  The number of hospital admissions
Healthcare usage | 3 months
  The healthcare usage expressed by the relevant medical assistance usage

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Bamidis, PhD, Principal Investigator — Associate Professor
Locations (2):
- Greece (2):
  - AHEPA University Hospital of Thessaloniki, Thessaloniki
  - Laboratory of Medical Physics, AUTH, Thessaloniki

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Cichosz SL, Ehlers LH, Hejlesen O. Health effectiveness and cost-effectiveness of telehealthcare for heart failure: study protocol for a randomized controlled trial. Trials. 2016 Dec 12;17(1):590. doi: 10.1186/s13063-016-1722-5. PMID 27955682
- [Derived] Billis A, Pandria N, Mouratoglou SA, Konstantinidis E, Bamidis P. Development of Cognitive and Physical Exercise Systems, Clinical Recordings, Large-Scale Data Analytics, and Virtual Coaching for Heart Failure Patients: Protocol for the BioTechCOACH-ForALL Project. JMIR Res Protoc. 2020 May 4;9(5):e17714. doi: 10.2196/17714. PMID 32364512